CLINICAL TRIAL: NCT06427915
Title: Studying GlucOse anD Appetite ResponseS With Alternatives to Pop (SODA-SWAP)
Brief Title: Studying Glucose and Appetite Response With Alternatives to Soda Pop
Acronym: SODA-SWAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olipop, PBC (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BIO-2401
Record Dates: First submitted 2024-05-16; First posted 2024-05-24 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Healthy Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soda consumption in fasted state (Experimental): One 12oz serving of soda consumed alone after a 4 hour fasting period
  Interventions: Other: OLIPOP prebiotic soda; Other: Traditional sugar-sweetened cola
- Soda consumption with a defined carbohydrate rich meal (Experimental): One 12oz serving of soda consumed with a defined carbohydrate rich meal after a 4 hour fasting period
  Interventions: Other: OLIPOP prebiotic soda; Other: Traditional sugar-sweetened cola

INTERVENTIONS:
Other: OLIPOP prebiotic soda — 12oz serving containing Carbonated Water, OLISMART(TM) (Cassava Root Fiber, Acacia Fiber, Guar Fiber, Nopal Cactus*, Marshmallow Root*, Calendula Flower*, Kudzu Root*), Cassava Root Syrup, Apple Juice Concentrate, Lime Juice, Natural Cola Flavor, Alpinia Galanga Root*, Stevia Leaf*, Himalayan Pink Salt, Green Tea Caffeine*, Natural Caramel Flavor, Natural Vanilla Flavor, Cinnamon* (*Extract)
Other: Traditional sugar-sweetened cola — 12oz serving containing carbonated water, high fructose corn syrup, caramel color, phosphoric acid, natural flavors, caffeine

SUMMARY:
The primary aim of this clinical trial is to determine the acute effects of OLIPOP (a lower sugar, high fiber prebiotic soda) consumption, compared to consumption of a commercially available sugar-sweetened soda pop, on blood glucose in response to the beverages alone and in combination with a carbohydrate-rich mixed lunch meal in free-living, generally healthy adults.This study will consist of one screening/randomization clinic visit (day 0) and one follow-up clinic visit (day 5), with participants consuming study products on their own (e.g., at home) following an assigned treatment sequence on days 1, 2, 3, and 4. The main questions answered by this trial are the impacts of a prebiotic rich soda versus a traditional soda on: 1) blood glucose levels with and without a meal, 2) perceived hunger levels, 3) perceived alertness levels and 4) total caloric intake.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥18 to ≤65 years of age at visit 1a.
2. Body mass index (BMI) of ≥25.0 kg/m2 to <35.0 kg/m2 at visit 1a.
3. Fasting capillary (fingerstick) glucose <126 mg/dL at visit 1a. One repeat will be allowed for glucose values between ≥126 and ≤140 mg/dL (same day if subjects are confirmed fasting or a separate day if subjects were not fasting). If a repeat is taken, the second reading will be used to determine eligibility.
4. Willing to wear a continuous glucose monitor (CGM) sensor throughout study period and willing to adhere to instructions/ restrictions associated with the proper use and care of the CGM.
5. Non-user or former user (cessation ≥12 months) of tobacco or nicotine products (e.g., cigarette smoking, vaping, chewing tobacco) with no plans to begin use during the study period.
6. Non-user of marijuana and hemp products, including cannabidiol (CBD) products, within 60 d of visit 1a.
7. Willing to avoid alcohol 24 h prior to visit 1a/1b and throughout the study.
8. Willing to maintain habitual diet (with the exception of study products) and physical activity patterns throughout the trial.
9. Willing to use personal smart phone with operating system (Android version 12.0 or newer; Apple iPhone operating system (iOS) version 16 or newer) capable of downloading the Dexcom G7 CGM app and the Cronometer app for diet records.
10. Willing to adhere to all study procedures and sign forms providing informed consent to participate in the study and authorization to release relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. Inability to consume a standard 12 fl. oz. carbonated beverage with or without food within 15 min.
2. Extreme dietary habits (e.g., Atkins diet, very high protein, and/or vegan) in the judgment of the Investigator or has been diagnosed with an eating disorder.
3. Habitual (e.g., daily) use of fiber supplements or prebiotic supplements within 30 d of visit 1a.
4. Known allergy or sensitivity to any of the ingredients in the study products and/or meals provided.
5. Weight loss or gain >4.5 kg within 90 d of visit 1a.
6. Currently or planning to be on a weight loss or weight gain/ muscle-building regimen program during the study.
7. Use of vitamin C-containing supplements (including multivitamins) within 24 hours of visit 1a and during the study intervention period.
8. Shift workers with eating patterns not consistent with the study product consumption schedule.
9. History or presence of uncontrolled and/or clinically important endocrine, cardiovascular, pulmonary, hepatic, renal, hematologic, immunologic, dermatologic, rheumatic, and/or biliary conditions that, in the opinion of the Principal Investigator, could interfere with the interpretation of the study results.
10. Uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the blood pressure measured at visit 1a.
11. Gastrointestinal condition that could potentially interfere with absorption of the study product (e.g., inflammatory bowel syndrome, inflammatory bowel disease (Crohn's or ulcerative colitis), celiac disease, history of gastric bypass surgery).
12. Use of oral or injectable steroids (topical and inhaled are allowed) within 90 d of visit 1a.
13. Use of products containing salicylic acid (skin-care products are allowed if not used on the area surrounding the CGM sensor) within 24 hours of visit 1a/1b and during the study intervention period. If use occurs during the intervention period (e.g., subject takes an aspirin), details of the use (e.g., time, amount, product) should be documented.
14. Unstable use of any prescription medications that affect blood glucose levels, whereby stable is defined as no change in regimen within 90 d prior to visit 1a. Examples include diabetes medications, glucagon-like-peptide-1 (GLP-1) agonists, medications for anxiety, attention deficit/hyperactivity disorder (ADHD), depression, and other mental health problems (e.g., clozapine, olanzapine, quetiapine, and risperidone), thyroid hormone replacement medications, statins, protease inhibitors, adrenergic receptor blockers, and isotretinoin.
15. History or presence of cancer, except non-melanoma skin cancer, within 2 years of visit 1a.
16. Exposure to any non-registered drug product or has participated in another intervention study within 30 d prior to visit 1a.
17. Signs or symptoms of an active infection of clinical relevance within 5 d of visit 1a. The visit may be rescheduled such that all signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 d prior to visit 1a.
18. Recent history (within 12 months of visit 1) of alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz. beer, 5 oz. wine, or 11⁄2 oz. distilled spirits).
19. History of any major trauma or major surgical event within 60 d of visit 1a.
20. Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source document.
21. Any condition the Investigator believes would interfere with his ability to provide informed consent, comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Blood Glucose iAUC | For 2 hours post intervention
  Incremental area under the curve (iAUC) for glucose from t = -30 min prior to test product consumption to t = 120 min following test-product consumption (iAUC0-120 min), where t = 0 is the start of beverage consumption either alone or in combination with a meal (depending on the test sequence).

SECONDARY OUTCOMES:
Blood Glucose Cmax | For 2 hours post intervention
  Blood glucose maximum concentration
Time to Blood Glucose Cmax (Tmax) | For 2 hours post intervention
  Time to maximum blood glucose concentration
Blood Glucose Rise 0-2 Hours | For 2 hours post intervention
  The maximum concentration above the average baseline glucose concentration within the 2-hour period following study product consumption, expressed as a percentage of the average baseline glucose concentration
Blood Glucose Dip 2-3 Hours | For time frame of 2 to 3 hours post intervention
  The difference between the lowest glucose concentration in hours 2-3 after study product consumption and the average baseline glucose concentration, expressed as a percentage of average baseline glucose concentration
Blood Glucose Reduction | For time frame of 2 to 3 hours post intervention
  The number of participants with a reduction in glucose in hours 2-3 after study product consumption compared to the average baseline glucose concentration
Time Until Next Meal | Within same day post interevention
  The number of minutes after consumption of the study product that elapsed before the next meal of at least 50 kcal is consumed
Energy Intake - Short Term | For time frame of 3 to 4 hours post intervention
  Energy intake (kcals) within 3 to 4 hours post-product consumption
Energy Intake - 24 Hours | Time frame from 4 hours before the participant's breakfast to 20 hours after participant's breakfast
  The total daily consumption covers the full period from 4 hours before the participant's breakfast to 20 hours after
Change in Perceived Hunger Level | For time frame of 2 to 3 hours post intervention
  The change in hunger ratings from pre-meal to post meal where post meal is defined as the average of the hunger ratings in the 2- 3 hour time frame
Change in Perceived Alertness Level | For time frame of 2 to 3 hours post intervention
  The change in alertness ratings from pre-meal to post meal where the post meal is defined as the average alertness ratings in the 2-3 hour time frame

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis, Addison, Illinois, United States